CLINICAL TRIAL: NCT00066118
Title: The Casa Pia Study of the Health Effects of Dental Amalgam in Children.
Brief Title: Health Effects of Silver-Mercury Dental Fillings
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Timothy DeRouen, Professor Emeritus of Oral Health Sciences, School of Dentistry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10085; U01DE011894 (NIH); 95-0401-A 13 (Other: UW Human Subjects Division); NIDCR-11894 (Other: NIDCR); NCT00000365 (obsolete NCT alias)
Record Dates: First submitted 2003-08-04; First posted 2003-08-05 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Caries, Dental
Keywords: neurologic; nerve conduction; neurobehavioral; renal disease
MeSH Terms: conditions — Dental Caries; Neurologic Manifestations; Kidney Diseases

INTERVENTIONS:
Device: Dental amalgam restorations

SUMMARY:
The purpose of this study is to determine whether there are detectable health effects of low-level mercury exposure (from normal exposure to mercury-containing dental fillings) in the known target organs/systems affected by elemental mercury exposure.

DETAILED DESCRIPTION:
The Casa Pia Study of the Health Effects of Dental Amalgam in Children is a randomized, prospective clinical trial with the overall goal of determining if there are detectable health effects due to exposure from mercury-containing dental amalgam fillings. Children, thought to be the population most susceptible to any possible health effects, were randomly assigned to one of two treatment groups (total n=507). Subjects were originally enrolled at ages between 8-10 years of age. To participate, subjects must have: Dental caries in at least one posterior tooth; no prior exposure to dental amalgam; a blood lead of <15ug/L; a urinary mercury level of <10ug/L; an IQ as measured by the CTONI of >67; and no prior or existing serious medical or neurologic condition. One group received only dental filling materials other than those containing mercury (plastic and ceramic composites), while the other group received mercury amalgam fillings where appropriate (in large restorations in back teeth), but the alternative materials everywhere else. Both treatment regimens are standard-of-care throughout the world. Subjects receive ongoing dental care via the study clinics, and continue to receive dental fillings as needed based on group assignment. The target organs of mercury exposure are renal and neurological. Baseline and annual repeated measures are taken on all subjects for renal function, nerve conduction velocity and a large battery of neurobehavioral tests. Follow-up is planned for a period of 7 years

ELIGIBILITY:
* Age 8-10 years of age
* Dental caries in at least one posterior tooth.
* No prior exposure to dental amalgam
* Blood lead of <15ug/L
* Urinary mercury level of <10ug/L
* IQ as measured by the CTONI of >67
* No prior or existing serious medical or neurologic condition

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 507
Dates: Start 1996-08; Primary Completion 2005-07 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Memory
Rey Auditory Verbal Learning,
Finger Windows,
Visual Learning
Visual Motor Functions
Drawing, MatchingP
Pegboard sub-tests from the Wide Range Assessment of Visual Motor Abilities.
Attention/Concentration
Coding
Symbol Search
Digit Span
Standard Reaction Time
Stroop
Trails A and B.
Neurological: Nerve Conduction Velocity

CONTACTS AND LOCATIONS:
Overall Officials: Timothy DeRouen, Principal Investigator — University of Washington; Michael Martin, Study Chair — University of Washington
Locations (1):
- University of Washington, School of Dentistry, Seattle, Washington, United States

REFERENCES:
- [Result] DeRouen TA, Martin MD, Leroux BG, Townes BD, Woods JS, Leitao J, Castro-Caldas A, Luis H, Bernardo M, Rosenbaum G, Martins IP. Neurobehavioral effects of dental amalgam in children: a randomized clinical trial. JAMA. 2006 Apr 19;295(15):1784-92. doi: 10.1001/jama.295.15.1784. PMID 16622140
- [Result] Bernardo M, Luis H, Martin MD, Leroux BG, Rue T, Leitao J, DeRouen TA. Survival and reasons for failure of amalgam versus composite posterior restorations placed in a randomized clinical trial. J Am Dent Assoc. 2007 Jun;138(6):775-83. doi: 10.14219/jada.archive.2007.0265. PMID 17545266
- [Result] Woods JS, Martin MD, Leroux BG, DeRouen TA, Leitao JG, Bernardo MF, Luis HS, Simmonds PL, Kushleika JV, Huang Y. The contribution of dental amalgam to urinary mercury excretion in children. Environ Health Perspect. 2007 Oct;115(10):1527-31. doi: 10.1289/ehp.10249. PMID 17938746
- [Result] Lauterbach M, Martins IP, Castro-Caldas A, Bernardo M, Luis H, Amaral H, Leitao J, Martin MD, Townes B, Rosenbaum G, Woods JS, Derouen T. Neurological outcomes in children with and without amalgam-related mercury exposure: seven years of longitudinal observations in a randomized trial. J Am Dent Assoc. 2008 Feb;139(2):138-45. doi: 10.14219/jada.archive.2008.0128. PMID 18245680
- [Result] Woods JS, Martin MD, Leroux BG, DeRouen TA, Bernardo MF, Luis HS, Leitao JG, Kushleika JV, Rue TC, Korpak AM. Biomarkers of kidney integrity in children and adolescents with dental amalgam mercury exposure: findings from the Casa Pia children's amalgam trial. Environ Res. 2008 Nov;108(3):393-9. doi: 10.1016/j.envres.2008.07.003. Epub 2008 Aug 21. PMID 18721920
- [Result] Woods JS, Martin MD, Leroux BG, DeRouen TA, Bernardo MF, Luis HS, Leitao JG, Simmonds PL, Echeverria D, Rue TC. Urinary porphyrin excretion in children with mercury amalgam treatment: findings from the Casa Pia Children's Dental Amalgam Trial. J Toxicol Environ Health A. 2009;72(14):891-6. doi: 10.1080/15287390902959557. PMID 19557617